CLINICAL TRIAL: NCT04047108
Title: pedCAPNETZ - Development and Detailed Characterization of a Cohort for Community Acquired Pneumonia (CAP) in Childhood and Adolescence
Brief Title: pedCAPNETZ - Community Acquired Pneumonia (CAP) in Childhood and Adolescence
Acronym: pedCAPNETZ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: pedCAPNETZ
Record Dates: First submitted 2019-05-16; First posted 2019-08-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Establishment of a study network and patient cohort for pediatric CAP

DETAILED DESCRIPTION:
The aim of the project is the development of a large pediatric CAP patient cohort based on the established pedCAPNETZ pilot cohort. The main objective is to improve knowledge on etiology, epidemiology, diagnosis and management of pediatric CAP in a developed country. pedCAPNETZ will enable the systematic and detailed characterization of pediatric CAP cases on an epidemiological, clinical and biological level.

ELIGIBILITY:
Inclusion Criteria:

* age < 18
* symptoms of an acute lower respiratory tract infection with radiological confirmed pneumonia via ultrasound or chest x-ray

Exclusion Criteria:

* hospitalization for any reason within the last 28 days
* congenital or acquired immunodeficiency
* concomitant respiratory disease with impaired mucociliary clearance such as cystic fibrosis, primary ciliary dyskinesia, tracheostomy or other severe lung disease including pulmonary tuberculosis, malignancy, and cytostatic therapy during past 28 days or neutropenia (< 1000/µl) or relevant immunosuppressive treatment

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: CAP patients age < 18
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-12-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with pediatric community acquired pneumonia (pedCAP) across all different levels of health care | 5 years
  To establish a multicenter national, prospective, observational and longitudinal pedCAP database and collaborative research network
Prevalence of pedCAP and etiologies (composite outcome measures) across all different levels of health care | 5 years
  * Etiology of pedCAP in Germany
  * Clinical presentation of pedCAP
  * Predictors of severe clinical course of pedCAP
  * Diagnostics employed in management of pedCAP
  * Microbiology and virology of pedCAP
  * Radiology of pedCAP
  * Comorbidity in patients with pedCAP
  * Treatment patterns of pedCAP

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No